CLINICAL TRIAL: NCT05356299
Title: Analysis of the Magnetic Tape Bandage on Respiratory Functional Effects in Patients After Extubation Failure a Quasi-experimental Randomized Clinical Trial.
Brief Title: Analysis of the Magnetic Tape Bandage on Respiratory Functional Effects.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Doctor Peset (Other)
Responsible Party: Principal Investigator, Héctor Hernández Garcés, Dr. Hector Hernández-Garcés, Hospital Universitario Doctor Peset
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 123/20
Record Dates: First submitted 2022-04-18; First posted 2022-05-02 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Airway Extubation
Keywords: Airway extubation failure; Magnetictape; Invasive mechanical ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MagneticTape group (Experimental): The Magnetic Tape bandage will be placed by the patient's care team and will be placed in the anterior superior part of each hemithorax, matching the large vessels and lymph nodes, in the posterior part of the thorax in the paravertebral area from C3 to T9 and in the subcostal region, following the direct innervation of the thorax and shoulder girdle, as well as the dorsal levels with lateral horns that control the vascularisation of the thorax and shoulder girdle.
  Interventions: Other: Magnetictape bandage application

INTERVENTIONS:
Other: Magnetictape bandage application — The Magnetic Tape bandage will be placed by the patient's care team and will be placed in the anterior superior part of each hemithorax, matching the large vessels and lymph nodes, in the posterior part of the thorax in the paravertebral area from C3 to T9 and in the subcostal region, following the direct innervation of the thorax and shoulder girdle, as well as the dorsal levels with lateral horns that control the vascularisation of the thorax and shoulder girdle.

SUMMARY:
Invasive mechanical ventilation (IMV) is the mainstay of supportive care in acute respiratory failure. However, maintaining ventilatory support beyond what is necessary may increase the risk of nosocomial infections, favour respiratory muscle atrophy, prolong ICU stay and increase hospital costs. Similarly, premature withdrawal of ventilatory support may increase ICU patient mortality by requiring reintubation. The MV weaning process is nothing more than the set of procedures that lead to the restoration of normal ventilation of the patient, freeing him/her from ventilatory support and eventually also from an artificial airway. This is a gradual process that can take a significant amount of hospitalisation time, so much so that it could even correspond to 40% of the entire period of ventilatory support. Currently, the process of disconnection from IMV is based on the performance of a spontaneous ventilation test (SVT) either with an unsupported oxygen source or with low ventilator support , with a duration of 30 to 120 minutes.

One of the causes that may condition the viability of SVT is respiratory muscle weakness, which may be ventilator-induced. This condition is a syndrome characterised by the appearance of diffuse and symmetrical muscle weakness affecting 26-65% of patients mechanically ventilated for more than 5 days. Muscle wasting has been demonstrated by ultrasonography with an 18% reduction in the cross-sectional area of the rectus femoris muscle on the 10th day of evolution. This syndrome is associated with an increase in mechanical ventilation time and a 2 to 5-fold increase in mortality. Based on the above, the assessment of respiratory muscle strength should form part of the disconnection protocols of our units. The most studied parameters that provide us with information on patient readiness to face this process are f/Vt, PIM and P(O.1). Recently, the study of the diaphragm by ultrasonography is becoming a valid alternative technique for the study of the state of the muscle most involved in spontaneous breathing.

DETAILED DESCRIPTION:
Invasive mechanical ventilation (IMV) is the mainstay of supportive care in acute respiratory failure. However, maintaining ventilatory support beyond what is necessary may increase the risk of nosocomial infections, favour respiratory muscle atrophy, prolong Intensive Care Units (ICU) stay and increase hospital costs. Similarly, premature withdrawal of ventilatory support may increase ICU patient mortality by requiring reintubation. The Mechanical Ventilation (MV) weaning process is nothing more than the set of procedures that lead to the restoration of normal ventilation of the patient, freeing him/her from ventilatory support and eventually also from an artificial airway. This is a gradual process that can take a significant amount of hospitalisation time, so much so that it could even correspond to 40% of the entire period of ventilatory support. Currently, the process of disconnection from IMV is based on the performance of a spontaneous ventilation test (SVT) either with an unsupported oxygen source or with low ventilator support , with a duration of 30 to 120 minutes.

One of the causes that may condition the viability of SVT is respiratory muscle weakness, which may be ventilator-induced. This condition is a syndrome characterised by the appearance of diffuse and symmetrical muscle weakness affecting 26-65% of patients mechanically ventilated for more than 5 days. Muscle wasting has been demonstrated by ultrasonography with an 18% reduction in the cross-sectional area of the rectus femoris muscle on the 10th day of evolution. In addition, this syndrome is associated with an increase in mechanical ventilation time and a 2 to 5-fold increase in mortality. Based on the above, the assessment of respiratory muscle strength should form part of the disconnection protocols of our units. The most studied parameters that provide us with information on patient readiness to face this process are f/Vt, Inspiratory Maximum Pressure (IMP) and Airway Occlusion Pressure P(O.1). Recently, the study of the diaphragm by ultrasonography is becoming a valid alternative technique for the study of the state of the muscle most involved in spontaneous breathing.

Magnetic Tape® is an elastic adhesive bandage with a longitudinal elongation of 50-60% designed to facilitate the process of metameric normalisation by producing physical ionisation when it comes into contact with electromagnetic fields such as those produced in the skin thanks to the formulation of cations (+ ions) and anions (- ions) that it incorporates per square centimetre, acting both polarities (positive and negative) indistinctly and uninterruptedly at the same time, painless and non-invasive, stimulating the cutaneous receptors and nerves, allowing neural stimulation. The electromagnetic field acts as the vehicle to induce the flow of ions (physical ionisation) and does not stimulate the nerve tissue itself as electrical stimulation does directly. However, once the ion flow is created, the mechanism of electrical and magnetic stimulation at the neural level is the same, producing depolarisation of the axon and initiation of the action potential.

The skin is the largest sensory organ in the body and is highly innervated. The nerve fibres it contains are the dendritic limbs of sensory neurons whose cell bodies are located in the dorsal root ganglia.

The main effects studied so far are: 1) It provides a considerable, significant and immediate change in the improvement of joint Range of Movement (ROM); 2) It produces a decrease or elimination of perceived pain in all phases of therapeutic action such as prevention, treatment, recovery, readaptation or performance; 3) It helps to normalise the autonomic nervous system; 4) It normalises the body's dermal temperature; 5) It helps to reduce the collection of liquid after a contusion or fall; 6) It helps to produce myo-normalisation either by relaxation or stimulation; 7) It helps to improve the symptoms caused by scar adhesions.

We consider it interesting, as a starting point in the field of medicine, to present this work and evaluate the effect of Magnetic Tape on the respiratory musculature and, therefore, on the parameters most commonly used for the evaluation of the same in ventilated patients who are going to undergo a Spontaneus Ventilation Test (SVT).

ELIGIBILITY:
Inclusion Criteria:

* All patients who have received IMV for more than 48 hours and are intended to start the ventilator weaning process.

Exclusion Criteria:

* Adequate oxygenation (SatO2>90% or PaO2>60mmHg, FiO2<0.4 and PEEP <7).
* Patients under deep sedation+/- muscle relaxation
* Patients in need of OTI due to structural alterations of the central nervous system
* Patients with a history of previously known neurological disease
* Patients with wounds or burns in the paravertebral region, interscapular or subcostal region
* Patients with active oncological disease
* Patients with contraindication for exposure to electromagnetic fields
* Patients under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Peak Inspiratory Pressure | 5 minutes, 24 hours
  The measurement will be performed using the ventilator software (Puritan Bennett 980 / 840, Medtronic, Dublin Ireland). Change from Baseline Peak Inspiratory Pressure at 24 h.

SECONDARY OUTCOMES:
Airway Occlusion Pressure | 5 minutes, 12 hours, 24 hours
  The measurement will be performed using the software and the ventilator curves (Puritan Bennett 980 / 840, Medtronic, Dublin Ireland).
Diaphragmatic excursion and Diaphragmatic thickening fraction | 5 minutes, 12 hours, 24 hours
  Assessment of diaphragmatic activity will be performed using ultrasound equipment.
Peak coughing flow | 5 minutes, 12 hours, 24 hours
  The measurement will be performed using the ventilator software (Puritan Bennett 980 / 840, Medtronic, Dublin Ireland).
Ph | 5 minutes, 12 hours, 24 hours
  Will be performed by analysis of arterial vs. venous blood sample.
PaCO2, PaO2 | 5 minutes, 12 hours, 24 hours
  Will be performed by analysis of arterial vs. venous blood sample.
Time of mechanical ventilation | 5 minutes, 12 hours, 24 hours
  The number of days the patient has been under OTI since intubation shall be recorded.
Weaning time | 5 minutes, 12 hours, 24 hours
  The number of days from the first PVE to extubation of the patient shall be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Hector Hernández-Garcés, PhD, Principal Investigator — University Hospital Dr. Peset
Locations (1):
- Hospital Universitario Doctor Peset, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Result] Esteban A, Alia I, Ibanez J, Benito S, Tobin MJ. Modes of mechanical ventilation and weaning. A national survey of Spanish hospitals. The Spanish Lung Failure Collaborative Group. Chest. 1994 Oct;106(4):1188-93. doi: 10.1378/chest.106.4.1188. PMID 7924494
- [Result] Esteban A, Ferguson ND, Meade MO, Frutos-Vivar F, Apezteguia C, Brochard L, Raymondos K, Nin N, Hurtado J, Tomicic V, Gonzalez M, Elizalde J, Nightingale P, Abroug F, Pelosi P, Arabi Y, Moreno R, Jibaja M, D'Empaire G, Sandi F, Matamis D, Montanez AM, Anzueto A; VENTILA Group. Evolution of mechanical ventilation in response to clinical research. Am J Respir Crit Care Med. 2008 Jan 15;177(2):170-7. doi: 10.1164/rccm.200706-893OC. Epub 2007 Oct 25. PMID 17962636
- [Result] Esteban A, Alia I, Tobin MJ, Gil A, Gordo F, Vallverdu I, Blanch L, Bonet A, Vazquez A, de Pablo R, Torres A, de La Cal MA, Macias S. Effect of spontaneous breathing trial duration on outcome of attempts to discontinue mechanical ventilation. Spanish Lung Failure Collaborative Group. Am J Respir Crit Care Med. 1999 Feb;159(2):512-8. doi: 10.1164/ajrccm.159.2.9803106. PMID 9927366
- [Result] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Result] De Jonghe B, Sharshar T, Lefaucheur JP, Authier FJ, Durand-Zaleski I, Boussarsar M, Cerf C, Renaud E, Mesrati F, Carlet J, Raphael JC, Outin H, Bastuji-Garin S; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Paresis acquired in the intensive care unit: a prospective multicenter study. JAMA. 2002 Dec 11;288(22):2859-67. doi: 10.1001/jama.288.22.2859. PMID 12472328
- [Result] Ali NA, O'Brien JM Jr, Hoffmann SP, Phillips G, Garland A, Finley JC, Almoosa K, Hejal R, Wolf KM, Lemeshow S, Connors AF Jr, Marsh CB; Midwest Critical Care Consortium. Acquired weakness, handgrip strength, and mortality in critically ill patients. Am J Respir Crit Care Med. 2008 Aug 1;178(3):261-8. doi: 10.1164/rccm.200712-1829OC. Epub 2008 May 29. PMID 18511703